CLINICAL TRIAL: NCT05015361
Title: Efficacy and Safety of Remimazolam Tosilate for Injection in Local Anesthesia Assisted Sedation -- a Multicenter, Randomized, Single Blind, Positive Drug Parallel Controlled Phase II Clinical Trial
Brief Title: A Trial of Efficacy and Safety of Remimazolam Tosilate for Injection in Local Anesthesia Assisted Sedation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR7056-204
Record Dates: First submitted 2021-08-11; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Local Anesthesia Assisted Sedation
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: Remimazolam Tosilate compared with Propofol Injection
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A/B (Experimental): Treatment group A: Remimazolam Tosilate Treatment group B: Remimazolam Tosilate
  Interventions: Drug: Remimazolam Tosilate
- Treatment group C (Active Comparator): Treatment group C: Propofol Injection.
  Interventions: Drug: Propofol Injection.

INTERVENTIONS:
Drug: Remimazolam Tosilate — Treatment group A: Remimazolam Tosilate; high dose Treatment group B: Remimazolam Tosilate; low dose
  Arms: Treatment group A/B
Drug: Propofol Injection. — Treatment group C: Propofol Injection.
  Arms: Treatment group C

SUMMARY:
To evaluate the efficacy and safety of Remimazolam Tosilate for injection in local anesthesia assisted sedation, and to explore the dose range of remazolam toluenesulfonate for injection in local anesthesia assisted sedation.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects requiring local anesthesia assisted sedation
3. Male or female
4. Meet the weight standard
5. Conform to the ASA Physical Status Classification

Exclusion Criteria:

1. Previous respiratory or pulmonary diseases
2. Subjects who had received general anesthesia
3. Subjects with a history of myocardial infarction or unstable angina pectoris
4. Subjects with atrioventricular block or cardiac insufficiency
5. Subjects with a history of ischemic stroke or transient ischemic attack
6. Subjects with poor blood pressure control after medication
7. Subjects with abnormal clotting function
8. Subjects with a history of mental illness and a history of cognitive impairment epilepsy
9. Subjects with a history or possibility of a difficult airway
10. Subject with a history of substance abuse and drug abuse
11. Abnormal values in the laboratory
12. Allergic to a drug ingredient or component
13. Pregnant or nursing women
14. No birth control during the specified period of time
15. Participated in clinical trials of other drugs (received experimental drugs)
16. The inestigators determined that other conditions were inappropriate for participation in this clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-07-04 (Actual)

PRIMARY OUTCOMES:
The time to maintain target sedation as a percentage of the total study administration time. | through study completion,an average of about 1 hour

SECONDARY OUTCOMES:
Proportion of subjects who achieved target sedation within 3 minutes after starting intravenous injection of load dose test drugs; | 3 minutes after administration
Proportion of subjects receiving remedial sedation; | through study completion,an average of about 1 hour
The time from the start of intravenous injection of load dose test drug to the first achievement of target sedation; | Time to achieve target sedation, an average of about 4 minutes
The time from stopping infusion of test drugs to reaching MOAA/S level 5 for the first time after operation | Recovery time, an average of about 7 minutes
Anesthesiologists' satisfaction with sedation | through study completion,an average of about 1 hour
Evaluation of subjects' satisfaction with sedation treatment; | through study completion,an average of about 1 hour
Incidence of anterograde amnesia. | through study completion,an average of about 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided